CLINICAL TRIAL: NCT07150546
Title: Combination External Radiation and 177Lu-DOTATATE for Large Gastrointestinal Neuroendocrine Tumors: A Single Arm Pilot Clinical Trial
Brief Title: Combination External Radiation and PRRT for Large GI Neuroendocrine Tumors.
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Pretesh Patel, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00008681; P30CA138292 (NIH); NCI-2025-05882 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00008681 (Other: Emory University Hospital/Winship Cancer Institute); RAD6422-24 (Other: Emory University Hospital/Winship Cancer Institute)
Record Dates: First submitted 2025-08-25; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Digestive System Neuroendocrine Tumor; Unresectable Digestive System Neuroendocrine Neoplasm; Unresectable Digestive System Neuroendocrine Tumor G1; Unresectable Digestive System Neuroendocrine Tumor G2
MeSH Terms: conditions — Gastro-enteropancreatic neuroendocrine tumor | interventions — Radiosurgery; lutetium Lu 177 dotatate; Lutetium; Lutetium-177; copper dotatate CU-64; Magnetic Resonance Spectroscopy; X-Rays; Ga(III)-DOTATOC; gallium Ga 68 dotatate; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Intervention Model Description: Pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (SBRT, 177Lu-DOTATATE) (Experimental): Patients undergo SBRT over 5 fractions in the absence of disease progression or unacceptable toxicity. Starting 4-10 weeks after completion of SBRT, patients receive SOC 177Lu-DOTATATE IV once every 8 weeks for 4 doses in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and/or MRI throughout the trial and undergo gallium Ga 68-DOTATATE PET/CT before treatment.
  Interventions: Radiation: Stereotactic Body Radiation Therapy; Drug: Lutetium Lu 177 Dotatate; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Radiation: Gallium Ga 68-DOTATATE; Procedure: Positron Emission Tomography; Other: Questionnaire Administration

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR, SBRT, SBRT, Stereotactic Ablative Body Radiation Therapy, stereotactic body radiation therapy
Drug: Lutetium Lu 177 Dotatate — Given IV
  Other Names: 177 Lu-DOTA-TATE, 177 Lu-DOTA-Tyr3-Octreotate, 177Lu-DOTA0-Tyr3-Octreotate, 437608-50-9, Lutathera, Lutetium (177Lu) Oxodotreotide; 177 Lu-DOTA-TATE, 177 Lu-DOTA-Tyr3-Octreotate, 177Lu-DOTA0-Tyr3-Octreotate, Lutathera, Lutetium (177Lu) Oxodotreotide, Lutetium Lu 177 DOTA(0)-Tyr(3)-Octreotate, Lutetium Lu 177 Dotatate; Lutetium Lu 177-DOTA-Tyr3-Octreotate,Lutetium Oxodotreotide Lu-177
Procedure: Computed Tomography — Undergo CT and PET/CT
  Other Names: CAT, CAT Scan, CAT scan, CAT Scan, Computed Axial Tomography, Computed Tomography, Computed Tomography, Computed Tomography, computed tomography, Computed Tomography, computerized axial tomography,; Computerized Axial Tomography, Computerized axial tomography (procedure), Computerized Tomography, computerized tomography, Computerized Tomography,; Computerized Tomography (CT) scan, CT, CT, CT, CT, CT SCAN, CT Scan, CT scan, CT Scan, CT Scan, CT Scan, CT Scan, tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance, Magnetic Resonance Imaging; Magnetic Resonance Imaging (MRI), Magnetic resonance imaging (procedure), Magnetic Resonance Imaging Scan, Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance, MR,MR Imaging, MRI; MRI Scan, MRIs, NMR Imaging, NMRI, Nuclear Magnetic Resonance Imaging, sMRI, Structural MRI
Radiation: Gallium Ga 68-DOTATATE — Undergo gallium Ga 68-DOTATATE PET/CT
  Other Names: (68)Ga-DOTA-TATE, 1027785-90-5, 68Ga-DOTA-0-Tyr3-Octreotate, 68Ga-DOTATATE, Gallium Ga 68 Oxodotreotide, GALLIUM OXODOTREOTIDE GA-68, Gallium-68 DOTA-DPhe1, Tyr3-octreotate
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography, PET, PET, Pet Scan, PET SCAN, PET scan, PET Scan, PET Scan, PET Scan, Positron Emission Tomography, Positron Emission Tomography,; Positron emission tomography (procedure), positron emission tomography scan, Positron Emission Tomography Scan, Positron-Emission Tomography, PT
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase I trial tests the safety and effectiveness of stereotactic body radiation therapy (SBRT) followed by 177Lu-DOTATATE peptide receptor radionuclide therapy (PRRT) in treating patients with large well-differentiated grade 1-2 digestive system neuroendocrine tumors that cannot be removed by surgery (unresectable). SBRT is a type of external radiation therapy that uses special equipment to position a patient and precisely deliver radiation to tumors in the body. The total dose of radiation is divided into smaller doses given over several days. This type of radiation therapy helps spare normal tissue. 177Lu-DOTATATE is a radioactive drug. It binds to a protein called somatostatin receptor, which is found on some neuroendocrine tumor cells. 177Lu-DOTATATE builds up in these cells and gives off radiation that may kill them. It is a type of radioconjugate and a type of somatostatin analog. Giving PRRT after SBRT may reduce the chances of the disease returning or getting worse, compared to the standard treatment of PRRT alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the rate of acute grade 3+ non-hematologic toxicity of PRRT after external radiation compared to historical control of PRRT alone.

SECONDARY OBJECTIVES:

I. To determine the rate of acute grade 2+ toxicity compared to historical control of PRRT alone.

II. To determine response rate of both large and small lesions at 3 months following treatment.

III. To determine progression free survival. IV. To describe patient-reported outcomes (PROs) of toxicity.

OUTLINE:

Patients undergo SBRT over 5 fractions in the absence of disease progression or unacceptable toxicity. Starting 4-10 weeks after completion of SBRT, patients receive standard of care (SOC) lutetium-177 DOTATATE (177Lu-DOTATATE) intravenously (IV) once every 8 weeks for 4 doses in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) and/or magnetic resonance imaging (MRI) throughout the trial and undergo gallium Ga 68-DOTATATE positron emission tomography (PET)/CT before treatment.

After completion of study treatment, patients are followed up at 90 days and then every 3 months for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age ≥ 18 years
* Patient must be able to provide study specific informed consent
* Pathologically confirmed neuroendocrine tumor fulfilling all of the following criteria
* Well-differentiated, grade 1-2
* Unresectable (prior resection is allowable), verified by tumor board or surgical oncology (surg onc)
* Progression after one or two prior lines of systemic therapy
* Somatostatin-receptor positive disease as determined by positive radiotracer-labeled DOTATATE PET/CT scan (modified Krenning score 3+)
* One or more large lesions measuring 3 or more cm on contrast-enhanced CT or MRI
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Estimated glomerular filtration rate (GFR) > 30 mL/min (within 90 days prior to study registration)
* Total bilirubin ≤ 3 x upper limit of normal (within 90 days prior to study registration)
* Albumin > 30 g/L (within 90 days prior to study registration)
* White blood cell (WBC) ≥ 2,000 cells/mm^3 (within 90 days prior to study registration)
* Platelets ≥ 70000 cells/mm^3 (within 90 days prior to study registration)
* Hemoglobin ≥ 8.0 g/dl (Note: The use of transfusion or other intervention to achieve hemoglobin [Hgb] ≥ 8.0 g/dl is acceptable.) (within 90 days prior to study registration)

Exclusion Criteria:

* Any prior radiation therapy including prior PRRT, external radiation, or Yttrium-90 radioembolization to the same site/region
* Contraindications to radiation therapy including inflammatory bowel disease, systemic sclerosis, etc.
* Brain metastases or any metastases extending into the spinal canal
* Unable to obtain confirmation of payment coverage for any planned radiation treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Acute Grade 3+ Non-Hematologic Adverse Events | Within 3 months of therapy
  Will evaluate acute grade 3+ non-hematologic toxicity (based on Common Terminology Criteria for Adverse Events version 5) compared to historical controls of peptide receptor radionuclide therapy alone. The list of non-hematologic acute grade 3+ treatment related adverse events will be summarized descriptively using frequencies and percentages of all captured toxicities by severity and relevance. An exact binomial test will then be used to compare the observed toxicity rate to the historical control rate, assessing if the observed rate significantly exceeds expected levels.

SECONDARY OUTCOMES:
Incidence of Acute Grade 2+ Non-Hematologic Adverse Events | Up to 12 months
  Non-hematologic acute grade 2+ treatment related adverse events will be summarized descriptively using frequencies and percentages of all captured toxicities by severity and relevance.
Response Rate | At 3 months
  The response rate based on Response Evaluation Criteria in Solid Tumors criteria of both large and small lesions at 3 months following treatment will be calculated along with 95% exact confidence intervals.
Progression Free Survival | At 12 months
  Progression free survival at 12 months will be estimated with the Kaplan-Meier method along with 95% confidence intervals.
Patient-Reported Health-Related Quality of Life | Up to 12 months
  Patient reported outcome will be summarized as mean, median, first quartile, third quartile, and standard deviation.

CONTACTS AND LOCATIONS:
Overall Officials: Pretesh Patel, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia